CLINICAL TRIAL: NCT04268108
Title: Clinical Study of Liquid Tumor Infiltrating Lymphocytes in Patients With Advanced Malignancies Resistance to Anti-PD-1 Therapy
Brief Title: L-TIL in Patients With Malignancy Resistance to Anti-PD-1 Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Liquid TIL
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-02

CONDITIONS: Advanced Solid Tumor
Keywords: liquid tumor-infiltrating lymphocytes; anti-PD-1; resistance; solid tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group 1: arm 1: secondary resistance to anti-PD-1 therapy: this patients group received liquid tumor infiltrating lymphocytes combined anti-PD-1 therapy.
  arm 2: primary resistance to anti-PD-1 therapy: this patients group received FC preconditioning before received liquid tumor infiltrating lymphocytes
  Interventions: Biological: liquid tumor infiltrating lymphocytes

INTERVENTIONS:
Biological: liquid tumor infiltrating lymphocytes — Isolatation and amplification PD-1+ cells from peripheral blood lymphocytes under GMP conditions for clinical use.

SUMMARY:
Safety and effectiveness of liquid tumor infiltrating lymphocytes in patients with advanced malignant tumors who have failed to anti-PD-1 therapy

ELIGIBILITY:
Inclusion Criteria:

* Expected lifespan is over 3 months
* malignant tumors diagnosed by pathological examination
* Imaging examination is at advanced stage with at least one measurable lesion
* Ineffective or resistant to previous anti-PD-1 therapy
* ECOG score 0-2
* Adequate organ function
* No other serious diseases that conflict with this protocol
* Women of childbearing age must check for a negative blood pregnancy test within 7 days, and subjects of childbearing age must use appropriate contraception during the test and within 3 months
* witten informed consent from the patients

Exclusion Criteria:

* Severe infectious disease within 4 weeks before enrollment
* Active hepatitis B or C virus or HIV infection
* Severe autoimmune disease or immunodeficiency disease
* Severe allergies
* Severe mental disorder
* Systematically used a large amount of glucocorticoids within 4 weeks before enrollment
* With severe heart, liver, kidney insufficiency, diabetes and other diseases
* Participation in other clinical studies in the past 3 months or having been treated with other gene products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2022-02-19 (Estimated); Study Completion 2022-06-19 (Estimated)

PRIMARY OUTCOMES:
the rate of reverse events | three months
  the rate of reverse events

SECONDARY OUTCOMES:
clinical benefit rate | three months
  the proportion of patients benefit from liquid tumor infiltrating lymphocytes
time to progression | six months
  from the date of therapy to the first date of determined progressive disease

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided
Need to solicit patients' consent whether to agree to share their information during the enrollment process,